CLINICAL TRIAL: NCT03838796
Title: A Prospective Cohort Study of the Effect of Lenvatinib Combined With TACE in Preventing the Recurrence in High-risk Patients With Hepatocellular Carcinoma
Brief Title: Lenvatinib Combined With TACE to Prevent the Recurrence in High-risk Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Director of the general surgery department, Huashan hospital, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huashan 004
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lenvatinib (Active Comparator): use lenvatinib after liver resection in HCC patients
  Interventions: Drug: lenvatinib
- lenvatinib and TACE (Active Comparator): use lenvatinib and TACE after liver resection in HCC patients
  Interventions: Drug: lenvatinib; Procedure: TACE

INTERVENTIONS:
Drug: lenvatinib — for patients <60kg, lenvatinib 8mg bid po for patients >60kg, lenvatinib 12mg bid po
  Other Names: lenvatinib treatment
Procedure: TACE — The patient underwent transfemoral hepatic artery angiography one month after surgery to observe whether there was tumor staining in the liver. If there was suspicious tumor staining, micro-catheter was superselected to the tumor blood vessel, the embolization agents and chemotherapy drugs were injected. If there was no tumor staining, a small amount of embolization agents were slowly injected into the artery.
  Other Names: transcatheter arterial chemoembolization
  Arms: lenvatinib and TACE

SUMMARY:
The purpose of the study is to observe the effect of Lenvatinib Combined With TACE in preventing the recurrence in high-risk patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Postoperative recurrence and metastasis of hepatocellular carcinoma(HCC）is the main problem during the treatment. Although with the development of medical science, some drugs have been found for the prevention and treatment of postoperative recurrence of HCC (such as postoperative application of interferon to prevent early tumor recurrence), but there is still no drug widely recognized.

Transcatheter arterial chemoembolization (TACE) is a palliative treatment for hepatocellular carcinoma. TACE can detect the early recurrence of tumor after liver resection, and has a complementary treatment effect on hidden residual lesions. For patients with high-risk, the tumor recurrence rate can be significantly reduced, and the tumor-free survival can be prolonged by TACE. Therefore, patients with high-risk of recurrence after resection were routinely arranged TACE treatment as an adjuvant treatment after surgery.

Lenvatinib is a multi-target receptor tyrosine kinase inhibitor (TKI), which mainly inhibits vascular endothelial growth factor(VEGF) receptor-1, 2, 3; fibroblast growth factors(FGF) receptor-1, 2, 3, 4; platelet derived growth factor receptor(PDGFR)α; RET and KIT, thereby inhibiting tumor cell proliferation, inducing apoptosis, and acting as an anti-angiogenesis. The REFLECT study showed that the median overall survival(OS) of the patients in the lenvatinib group was 13.6 months (95% CI, 12.1-14.9) and that in the sorafenib group was 12.3 months (95% CI, 10.4-13.9) , which reached a non-inferiority end point (HR = 0.92; 95% CI, 0.79-1.06). In addition, all secondary endpoints in the lenvatinib group were significantly better than the sorafenib group. A subgroup analysis based on Chinese patients showed that the OS of Lenvatinib was significantly 4.8 months longer than sorafenib group (15.0 months vs 10.2 months). Other three secondary endpoints, progression-free survival(PFS) (9.2 months vs 3.6) and time to progression(TTP)(11.0 months vs 3.7 months) and objective response rate(ORR) (21.5% vs 8.3%), were also significantly better in Lenvatinib group. Based on the above datas, lenvatinib will become a new choice for Chinese patients with HCC. It has also been approved by the FDA and CFDA as the first-line treatment for patients with advanced HCC.

So, this study is to observe the effect of lenvatinib combined with TACE in preventing the recurrence in high-risk patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* The characteristics of the treatment history:

No lenvatinib treatment history, no sorafenib allergies.

* The characteristics of the tumor:

The pathological results is hepatocellular carcinoma.

Meet any of the following articles:

Pathological prompt microvascular invasion(MVI) class II, and incorporate any of the following:Tumor number≥3,Tumor size≥8cm,Tumor margin is not clear and no complete capsule.

With the embolus in Portal vein, hepatic vein or bile duct. Preoperative rupture or invasion the adjacent organs.

* The characteristics of the patients:

The patient age was between 18-75. The American Society of Anesthesiologists(ASA）score was I-III. The Child-pugh score was A. Total bilirubin≤3.0 mg/dL, albumin≥28 g/L, AST, ALT, ALP≤5 times the upper limit of normal value.

Routine blood test: the neutrophil≥1.5×10^9/L, Hb≥8.5g/L，PLT≥75×10^9/L. The INR≤2.3. The Eastern Cooperative Oncology Group(ECOG) score was less than 2 points

Exclusion Criteria:

* R1/2 or palliative rescted tumor
* Pregnant or lactating women.
* Patients with other malignant tumor.
* Patients with mental illness.
* Patients participated in other clinical trials in last three months.
* Residual lesions showed by Postoperative digital subtraction angiography(DSA).
* Postoperative patients treated with other targeted drugs, PD1 antibody and other immunotherapies, FOLFOX systemic chemotherapy, and HuaiErKeLi drug treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years
  the survival time after liver resection without tumor recurrence or metastasis

SECONDARY OUTCOMES:
Overall survival | 5 years
  the survival time after liver resection

CONTACTS AND LOCATIONS:
Overall Officials: Lunxiu Qin, MD, Principal Investigator — Department of general surgery, Huashan hospital, Fudan University
Locations (1):
- Huashan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Llovet JM, Burroughs A, Bruix J. Hepatocellular carcinoma. Lancet. 2003 Dec 6;362(9399):1907-17. doi: 10.1016/S0140-6736(03)14964-1. PMID 14667750
- [Result] Sun HC, Tang ZY, Wang L, Qin LX, Ma ZC, Ye QH, Zhang BH, Qian YB, Wu ZQ, Fan J, Zhou XD, Zhou J, Qiu SJ, Shen YF. Postoperative interferon alpha treatment postponed recurrence and improved overall survival in patients after curative resection of HBV-related hepatocellular carcinoma: a randomized clinical trial. J Cancer Res Clin Oncol. 2006 Jul;132(7):458-65. doi: 10.1007/s00432-006-0091-y. Epub 2006 Mar 24. PMID 16557381
- [Result] Wang Z, Ren Z, Chen Y, Hu J, Yang G, Yu L, Yang X, Huang A, Zhang X, Zhou S, Sun H, Wang Y, Ge N, Xu X, Tang Z, Lau W, Fan J, Wang J, Zhou J. Adjuvant Transarterial Chemoembolization for HBV-Related Hepatocellular Carcinoma After Resection: A Randomized Controlled Study. Clin Cancer Res. 2018 May 1;24(9):2074-2081. doi: 10.1158/1078-0432.CCR-17-2899. Epub 2018 Feb 2. PMID 29420221
- [Result] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Derived] Chen JH, Lu L, Zhang XY, Xiang BD, Xu X, Li XC, Huang ZY, Wen TF, Luo LP, Huang J, Zhong JH, Liu ZK, Li CX, Long X, Zhu WW, Yang X, Wang CQ, Jia HL, Zhang JB, Zeng YY, Lu CD, Qin LX. Adjuvant lenvatinib in combination with transarterial chemoembolization for hepatocellular carcinoma patients with high risk of postoperative recurrence: A multicenter prospective cohort study. Hepatobiliary Pancreat Dis Int. 2025 Jun;24(3):277-285. doi: 10.1016/j.hbpd.2025.03.001. Epub 2025 Mar 26. PMID 40187927